CLINICAL TRIAL: NCT05199506
Title: A Single Center Prospective Study to Evaluate the Safety and Effectiveness of the Soliton® Rapid Acoustic Pulse (RAP)™Device for the Improvement in the Appearance of Cellulite.
Brief Title: Study to Evaluate the Safety and Effectiveness of the RAP Device for the Improvement in the Appearance of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02
Record Dates: First submitted 2021-11-22; First posted 2022-01-20 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Each leg/buttock will be treated with the RAP device (Experimental): Each leg will be treated with standard RAP treatment settings.One leg will receive treatments with 100Hz and the other with 50hz
  Interventions: Device: RAP

INTERVENTIONS:
Device: RAP — Treatment of cellulite with RAP device

SUMMARY:
The purpose of this single site clinical study is to evaluate the safety and effectiveness of the Soliton Rapid Acoustic Pulse (RAP) device for the improvement of cellulite comparing two different RAP treatment doses.

DETAILED DESCRIPTION:
This is a non-significant risk, single-center, prospective trial for safety, and efficacy using Soliton's RAP device for the improvement in the appearance of cellulite performed at 1 (one) clinical research site in the United States.

Approximately 15 healthy female participants between the age of 18-55 inclusive will be enrolled in this study.

Participants who sign the informed consent form and meet all the eligible criteria will be enrolled in the study. Each participant will undergo acoustic rapid pulse (RAP) treatments on each of the participants buttocks and legs. The participant's right buttock and leg will receive 100 Hz doses, and the participants left buttock and leg will receive 50 Hz doses.

Total study duration is anticipated to be at or less than 55 weeks from the first participant visit to the last participant observation visit. A total of 3 visits, plus two optional visits are planned for this study as listed below:

* Visit 1: Baseline/Screening (-30 Days to Day 0)
* Visit 2: Treatment (Day 0)
* Visit 3: 12-week Follow-Up Visit (+/- 14 Days)
* Visit 4: 26-week Follow-Up Visit (+/- 14 Days) (Optional)
* Visit 5: 52 Week Follow-Up Visit (+/- 14 Days) (Optional)

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment of cellulite in the thigh and/or buttock areas
* Area of moderate to severe cellulite on thigh and/or buttock for both legs using the Cellulite Dimple - At Rest Scale at Baseline with grades of 2 or 3 based on review of photos taken under the same lightening conditions planned for the trial.
* Body Mass Index (B.M.I.) is ≤ 30
* Participant will not have had invasive or energy-based cellulite treatments (liposuction, subcision, RF, laser, ESWT, etc.) for the prior 12 months.
* Participant will not have used topical based cellulite treatments for prior 6 months and will not use during the trial.
* Participant will not have used spray-on tanning treatments for 6 months prior to the initiation of the trial. Furthermore, participants will not use spray-on tanning treatments during the term of the trial.
* Participants must be able to provide written informed consent, understand and is willing to comply with all study related procedures and follow-up visits.

Exclusion Criteria:

* Participant is unwilling to have research photos taken of treatment areas in the presence of Sponsor's researchers.
* Participant is unwilling to have RAP treatment provided in the presence of Sponsor's researchers.
* Participant is pregnant or planning to become pregnant during the duration of the study.
* Participant is unwilling to commit to follow-up visits
* Metal or plastic implants in the area of the treatment (vascular stent, or implants in the hips, knees, etc.).
* Active electronic implants such as pacemakers, defibrillators.
* History of coagulopathy(ies) and/or on anticoagulant medication.
* Skin disorders (skin infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
* Any surgical procedure in the treatment areas in the prior 3 months or planned during the duration of the study.
* Participant is a current smoker.
* Participant has tattoo in treatment area.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Assessing safety | Immediately post treatment
  The primary safety short-term endpoint to be met if all treated participants were free from unexpected adverse events (UAEs) or serious adverse events (SAEs) attributable to the RAP treatment immediately post-treatment
Assessing safety | 12 weeks post treatment
  The primary safety short-term endpoint to be met if all treated participants were free from unexpected adverse events (UAEs) or serious adverse events (SAEs) attributable to the RAP treatment at the short-term (12-week) visit.
Assessing Efficacy | At 12 week follow up visit
  The primary effectiveness objective was to demonstrate improvement in the appearance of cellulite from the 100 Hz treatment is comparable to the 50 Hz treatment. Efficacy determined by the results of a blinded independent physician assessment (IPA) panel correctly identifying the 12-week post-treatment photographs from randomly placed side-by-side comparison of before and after photographs for both treatments. The primary effectiveness endpoint will be met if the rate of correctly identified before and after photos for 100 Hz treatment is not significantly lower than the 50 Hz treatment assessment.

SECONDARY OUTCOMES:
Assessing Participant Satisfaction | At the 12 week follow up visit
  Improvement in cellulite as measured by the percentage of participants who agree or strongly agree that the final photograph of the treatment area as compared to the baseline photograph, appears improved.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Capelli, MD, Study Director — Sponsor GmbH
Locations (1):
- The Practice of Brian Biesman, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Biesman BS, Capelli CC. Comparing safety and efficacy of acoustic subcision at two different rapid acoustic pulse rates to improve the appearance of cellulite. Lasers Surg Med. 2024 Jan;56(1):32-38. doi: 10.1002/lsm.23718. Epub 2023 Sep 11. PMID 37694399